CLINICAL TRIAL: NCT00215033
Title: Relationship Between Quantitative Epstein-Bar Viral(EBV) Titres and Post-Transplant Lymphoproliferative Disease
Brief Title: Relationship Between EBV and PTLD
Status: Terminated | Type: Observational
Why Stopped: sufficient data gathered to support conclusion
Sponsor: Children's Healthcare of Atlanta (Other)
Other Study IDs: 05-089
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2007-05

CONDITIONS: Pediatric Heart Transplant
Keywords: Epstein-Barr virus; pediatric health; cardiac; heart transplant; lymphoproliferative disease; post-transplant; pediatric transplant
MeSH Terms: conditions — Epstein-Barr Virus Infections; Lymphoproliferative Disorders

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the significance of an elevated quantitative EBV PCR and to determine the relationship between a EBV PCR value and the risk of developing PTLD.

DETAILED DESCRIPTION:
The relationship between Epstein-Barr virus and lymphoproliferative disease has been established, particularly in the immuno-suppressed patient. Over the past several years a quantitative EBV PCR lab test has been established. Unfortunately, the significance of an elevated test remains unclear. The relationship of a particular EBV PCR value and the risk of developing PTLD is unknown. The primary aims will be to determine the significance of an elevated quantitative EBV PCR and to determine the relationship between a EBV PCR value and the risk of developing PTLD. The study will be conducted through a retrospective chart review of approximately 160 patients and we will look at postoperative data including Quantitative EBV PCR results, the presence / absence of PTLD and the treatment of PTLD and results of EBV PCR with treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients undergone pediatric heart transplant
* followed by pediatric heart transplant program

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergone pediatric heart transplant
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2005-04; Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kogon, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States